CLINICAL TRIAL: NCT05313555
Title: The Effect of Violet Device Dosed UV-C Exposure on Healthy Hand Skin
Brief Title: The Effect of Violet Device Dosed Ultra Violet-C Light (UV-C) Exposure on Healthy Hand Skin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Archimedes Innovations, Pbc (Unknown)
Responsible Party: Principal Investigator, Gary Fisher, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00198624
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: ultraviolet light; light skin; skin changes; healthy volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ultraviolet lights (UV-B) (Active Comparator)
  Interventions: Device: Ultraviolet Light (UV-B)
- Ultraviolet lights (UV-C) (Experimental)
  Interventions: Device: Ultraviolet lights (UV-C)

INTERVENTIONS:
Device: Ultraviolet Light (UV-B) — This control group will receive a UV-B exposure as a positive control. Participants will have punch biopsies after exposure.
  Arms: Ultraviolet lights (UV-B)
Device: Ultraviolet lights (UV-C) — Violet is tabletop device that emits filtered UV-C (200nm-230nm; peak at 222nm). Participants will choose, based on availability, to be in groups that deliver 1 cycle, 10 cycles, 15 cycles or 25 cycles of the Violet. The subject will be exposed for no more than 5 minutes and 20 seconds in total. Participants will have punch biopsies after exposure.
  Other Names: Violet UV-C Light; Care222
  Arms: Ultraviolet lights (UV-C)

SUMMARY:
The purpose of this trial is to determine the safety of ultraviolet light (UV-C) irradiation as a method to sanitize hands instead of chemical-based sanitizers.

Eligible participants will be enrolled and receive treatment with the Violet UV-C device or UV-B. Punch biopsies will be performed following UV exposure to quantify any changes in cellular and molecular properties of the tissue.

ELIGIBILITY:
Inclusion Criteria

* Good general health
* Type 1 or type 2 skin (lightly colored skin)
* No history of skin disorders, disease states or physical conditions which would impair evaluation of the test sites
* Willingness and ability to follow the protocol
* No use of lotion or hand sanitizer 3 hours before the experiment

Exclusion Criteria:

* Has received an experimental drug or used an experimental device in the 30 days prior to admission to the study
* Undergoing treatment or taking medication that increases sun sensitivity
* History of keloids
* History of sensitivity to lidocaine or epinephrine
* Pregnant or nursing women, pregnancy status will be self-reported, women unsure of their pregnancy status will be excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Deoxyribonucleic acid (DNA) damage in the form of DNA base pair dimers measured by immunohistochemistry microscopy with statistical analysis. | Day 1 (visit 1 after light therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fisher, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No